CLINICAL TRIAL: NCT00285766
Title: A Phase III, Open-Label Study of the Safety, Tolerability and Efficacy of the Selegiline Transdermal System in Elderly Subjects With Major Depression
Brief Title: Safety, Tolerability and Efficacy of the Transdermal System in Elderly Subjects With Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Somerset Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S9303-P0204
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Major Depression
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: Selegiline Transdermal System

SUMMARY:
Objective of this 16-week, open-label study is to assess the safety and tolerability of once daily application of three doses of STS during continuous dosing in the treatment of elderly subjects with major depression. Subjects will have study visits (clinic visits) at beginning of study (baseline) and study weeks 1, 3, 5, 8, 12, and 16.

ELIGIBILITY:
* Men/Women in good health 65 years or older
* Ability to read, understand and sign study informed consent
* Major depression- mild to severe based on rating scale

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300
Dates: Start 2002-08; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Mohammed Bari, M.D., Chula Vista, California
  - Charles Meredith, M.D., San Diego, California
  - Daniel Zimbroff, M.D., Upland, California
  - Kathleen Toups, M.D., Walnut Creek, California
  - Abbey Strauss, M.D., Boynton Beach, Florida
  - Barry Baumel, M.D., Miami Beach, Florida
  - Margarita Nunez, M.D., St. Petersburg, Florida
  - Mildred Farmer, M.D., St. Petersburg, Florida
  - Larry Eisner, M.D., Tamarack, Florida
  - Andrew Cutler, M.D., Winter Park, Florida
  - Robert Riesenberg, M.D., Atlanta, Georgia
  - James Hartford, M.D., Florence, Kentucky
  - Mitchel Kling, M.D., Baltimore, Maryland
  - Louise Beckett, M.D., Oklahoma City, Oklahoma
  - Penny Barnhart, M.D., Wichita Falls, Texas